CLINICAL TRIAL: NCT04347161
Title: Implementation Strategies for Monitoring Adherence in Real Time
Acronym: iSMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Lung Cancer Research Foundation (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Katharine Rendle, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UPCC 20520; 834713 (Other: UPenn IRB)
Record Dates: First submitted 2020-04-01; First posted 2020-04-15 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer; Medication Adherence; Symptoms and Signs
Keywords: medication adherence; symptom management; non-small cell lung cancer; implementation science; digital health; behavioral science
MeSH Terms: conditions — Lung Neoplasms; Medication Adherence; Signs and Symptoms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Patients with lung cancer receiving oral targeted therapies at recruitment sites will be randomized (1:1 stratified by drug class and prescription status) to receive intervention or usual care.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and their care providers (including investigators) will not be blinded. The primary analyst and outcomes assessor will be blinded. Blinding may be broken in an emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Arm (Experimental): Participants in the intervention arm will be tracked and able to engage with the intervention (conversational agent) on their mobile telephone for 12 weeks.
  Interventions: Device: Conversational Agent/Chatbot
- Control Arm (Active Comparator): Patients in the control arm will receive usual care, which includes clinician-driven education on medication management and self-monitoring of symptoms.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Conversational Agent/Chatbot — Via text messages, the bidirectional, conversation agent provides specific dosing instructions and motivational reminders to promote oral targeted therapy adherence and symptom management. Patients can report symptoms at any time via text message and are also prompted to report symptoms and medication adherence at periodic intervals. Reported symptoms are monitored and managed algorithmically according severity. High-grade symptoms are triaged directly to the patients' cancer care team. Patients in the intervention arm will use MEMS caps to enable capture of the primary outcome and asked to complete longitudinal surveys.
  Arms: Intervention Arm
Other: Usual Care — Patients in the control arm will receive usual care, which includes receiving information about dosing and self-administration of oral therapy, and anticipatory guidance for patients regarding management of side effects. Patients in the control arm will use MEMS caps to enable capture of the primary outcome and asked to complete longitudinal surveys.
  Arms: Control Arm

SUMMARY:
The objective of this project is to identify effective strategies to help patients with lung cancer manage side effects and achieve optimal adherence to oral targeted therapies. To achieve this objective, we will evaluate the effect of a novel, bidirectional conversational agent, compared to usual care, on adherence to oral targeted therapies using a two-arm randomized controlled trial, and explore how multilevel factors impact the acceptability and effectiveness of this strategy by collecting qualitative and quantitative data from clinicians and patients.

DETAILED DESCRIPTION:
Drawing from insights in behavioral economics and implementation science, the goal of our project is to identify effective strategies for improving lung cancer outcomes by helping patients to better manage symptoms and adhere to oral therapies. Given the rapid increase in FDA-approved targeted therapies, the need for such strategies will continue to grow. Our central hypothesis is that conversational agent will improve adherence to oral therapies by targeting patient-level determinants of behavior change. The specific aims are to: 1) Test the effects of a patient-directed intervention (conversational agent) to improve adherence to oral targeted therapies in patients with non-small cell lung cancer.; and 2) Use mixed-methods approaches with clinicians and patients to explore multilevel factors shaping the acceptability, effectiveness, and future implementation of intervention into routine cancer care. Primary trial outcomes (adherence and persistence) will be measured using microelectronic monitoring system (MEMS) caps. Secondary outcomes will be assessed using longitudinal surveys and medical record data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18 years) with NSCLC at UPHS who is receiving one of the following nine oral therapies: afatinib, erlotinib, dacomitinib, gefitinib, osimertinib, alectinib, brigatinib, crizotinib, or lorlatinib.
* Patient possession of a mobile device that can send/receive SMS texts
* Ability to respond to questions and engage with "Penny" in English
* Ability to provide informed consent to participate in the study
* Approval from the patient's medical oncologist to be approached

Exclusion Criteria:

* Inability to respond to questions and engage with "Penny" in English
* Inability or unwillingness to provide informed consent to participate in the study
* Inability to engage with SMS text-messaging platform
* Concurrent enrollment in a therapeutic clinical trial
* Taking more than one oral targeted therapy or concurrent chemotherapy during the study window
* Lack of approval from the patient's oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2025-10-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine A Rendle, PhD,MSW,MPH, Principal Investigator — University of Pennsylvania; Samuel U Takvorian, MD, MSHP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Conversational Agent/Chatbot (Intervention): Participants in the intervention arm will be tracked and able to engage with the intervention (conversational agent) on their mobile telephone for 12 weeks.
  Conversational Agent/Chatbot: Via text messages, the bidirectional, conversation agent provides specific dosing instructions and motivational reminders to promote oral targeted therapy adherence and symptom management. Patients can report symptoms at any time via text message and are also prompted to report symptoms and medication adherence at periodic intervals. Reported symptoms are monitored and managed algorithmically according severity. High-grade symptoms are triaged directly to the patients' cancer care team. Patients in the intervention arm will use MEMS caps to enable capture of the primary outcome and asked to complete longitudinal surveys.
- Usual Care (Control): Patients in the control arm will receive usual care, which includes clinician-driven education on medication management and self-monitoring of symptoms.
  Usual Care: Patients in the control arm will receive usual care, which includes receiving information about dosing and self-administration of oral therapy, and anticipatory guidance for patients regarding management of side effects. Patients in the control arm will use MEMS caps to enable capture of the primary outcome and asked to complete longitudinal surveys.
Period: Overall Study
Arm/Group | Conversational Agent/Chatbot (Intervention) | Usual Care (Control)
Started | 38 | 37
Completed | 36 | 33
Not Completed | 2 | 4
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — No longer on study medication | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 20 | 34
  >=65 years | 24 | 17 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (2.4) | 61.3 (2.0) | 62.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 16 | 11 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Defined as number of patients who have 95% or greater adherent days across the study period based on their prescribed dose. Adherence data will be assessed via MEMS caps, which capture a date and time stamp each time the pill bottle is opened.
Time Frame: 12 weeks after study initiation or at therapy discontinuation, whichever is shorter
Population: Analysis population includes those patients with available adherence data (i.e., MEMS data successfully assessed).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 33 | 33
Participants | 18 | 20

2. Secondary Outcome: Persistence
Description: Defined as the average number of total days on the regimen before discontinuation measured using MEMS caps across participants
Time Frame: 12 weeks after study initiation or at therapy discontinuation, whichever is shorter
Measure: Mean (Standard Error); unit: days
Arm/Group | Conversational Agent/Chatbot (Intervention) | Usual Care (Control)
Number analyzed (Participants) | 33 | 33
days | 78.4 (2.3) | 79.8 (2.7)

ADVERSE EVENTS:
Time Frame: 12 week study duration
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/38 | 2/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 1/38 | 0/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=38) | Control Arm (N=37)
Discomfort using technology (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT04347161/Prot_SAP_000.pdf